CLINICAL TRIAL: NCT05657665
Title: Skin Tone Measurement Method Investigation for Pulse Oximetry
Status: Completed | Type: Observational
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Sponsor
Other Study IDs: ICBE-S-000880
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Skin Types; Pulse Oximetry
Keywords: Skin types; Pulse oximetry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational measurements of skin tone — Objective and subjective skin tone measurements will be performed.

SUMMARY:
The primary objective is to gather missing information in order to form a well-founded recommendation on which is the preferred skin pigmentation measurement (PPM) methods in the context of pulse-oximetry.

DETAILED DESCRIPTION:
Skin tone bias in pulse-oximetry (SpO2) needs to be addressed urgently. While skin pigmentation is a prime candidate for the root cause of skin tone bias in SpO2, more research is needed. F A solid comparison and recommendation requires evaluation of several additional aspects that affect accuracy, precision, and reproducibility of the PMMs.

Briefly, these additional aspects that are evaluated in this study are listed below:

* operator bias
* impact of operator color blindness
* probe pressure
* probe aperture size
* device stability
* impact of blood on pigmentation measurement
* feasibility of skin tone measurement on sides of fingers
* intra-operator variability

PMMs included in this study are:

Subjective color matching methods by using:

1. Von Luschan color scale
2. Fitzpatrick color scale
3. Pantone color scale

Objective probe-based measurements by using:

1. Konica Minolta CM700d (reflectance spectrometer)
2. Mx18 (erythema-melanin meter)
3. SPA99 (erythema-melanin meter)

Measurements will be performed on 5 relatively light skinned, and 5 relatively dark skinned volunteers (N=10 in total*). The study will be executed on the High-Tech Campus Eindhoven (Netherlands) and each participant will have 3 visits of approximately 1.5 to 2 hours/visit.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18-65 years)
2. Fluent in either English or Dutch
3. Participants who are willing and able to provide informed consent themselves.
4. People with Von Luschan scores <18 ('light skin' group) or > 25 ('dark skin' group).

Exclusion Criteria:

1. Skin conditions that could potentially interfere with the measurements:

   * piercings/ink/henna tattoos that cover the left forearm, hands, fingers or forehead
   * vascular or pigmentary or renal psoriasis
   * epidermal bullosum
   * other diseases that affect the skin (tone) of the body
2. COVID-19 exclusion criteria*:

   * Currently displaying COVID-19-related symptoms, namely a fever, cough and/or difficulty breathing
   * Having been positively tested as infected with COVID-19 in the past 14 days
   * Travelled to or from high risk COVID-19 areas in the past 14 days
   * Been in contact with a (suspected) COVID-infected person in the past 14 days
3. Not being able to travel to Eindhoven 3 times, and/or not being able to comply with the study procedures
4. Sunbathing during the study duration or substantial sun exposure (due to holidays for example).
5. Known allergic reaction to facial make-up
6. Usage of tanning sprays/cremes
7. Wearing make-up during the study visits (mascara is allowed)

   * No testing will be performed in the study. Participants will be asked if they have been positively tested.

Ages: 18 Years to 66 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers with Von Luschan scores <18 ('light skin' group) or > 25 ('dark skin' group.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Preferred skin PMM in the context of pulse-oximetry. | 10 months
  The primary objective is to complement a previous skin pigmentation study executed by Philips to gather missing information in order to form a well-founded recommendation on which is the preferred skin PPM in the context of pulse-oximetry.

CONTACTS AND LOCATIONS:
Locations (1):
- High Tech Campus, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: No
The plan is to perform data analysis by Philips Research. Thereafter data will be shared (de-identified) in a seperate publication that can be accessed overall.